CLINICAL TRIAL: NCT05320887
Title: The Impact of Cigarette Nicotine Content, E-Cigarette Nicotine Content and E-Cigarette Flavoring on Smoking Behavior in an Electronic Tobacco Marketplace
Brief Title: Cigarette and E-cigarette Nicotine Content in an Electronic Tobacco Marketplace (ETM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00080010; 5U54DA031659-09 (NIH)
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-03

CONDITIONS: Tobacco Use
Keywords: Cigarette smoking
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either low nicotine or normal nicotine content vaping devices with tobacco flavors only available
Who Masked: Participant
Masking Description: Participants are told their shopping trips are randomly selected, when they are actually being randomly selected between the two marketplace groups where only one flavor of e-liquid is available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal Nicotine Content Vape with all flavor e-liquids (Experimental): Normal Nicotine Content Vape with all flavor e-liquids
  Interventions: Other: Normal Nicotine Content Vape with all flavor e-liquids
- Normal nicotine content vape with tobacco e-liquids (Experimental): Normal nicotine content vape with tobacco e-liquids
  Interventions: Other: Normal nicotine content vape with tobacco e-liquids
- Low nicotine content vape with all flavor e-liquids (Experimental): Low nicotine content vape with all flavor e-liquids
  Interventions: Other: Low nicotine content vape with all flavor e-liquids
- Low nicotine content vape with tobacco e-liquids (Experimental): Low nicotine content vape with tobacco e-liquids
  Interventions: Other: Low nicotine content vape with tobacco e-liquids

INTERVENTIONS:
Other: Normal Nicotine Content Vape with all flavor e-liquids — Participants are randomly assigned to the order of each marketplace Group
  Arms: Normal Nicotine Content Vape with all flavor e-liquids
Other: Normal nicotine content vape with tobacco e-liquids — Participants are randomly assigned to the order of each marketplace Group
  Arms: Normal nicotine content vape with tobacco e-liquids
Other: Low nicotine content vape with all flavor e-liquids — Participants are randomly assigned to the order of each marketplace Group
  Arms: Low nicotine content vape with all flavor e-liquids
Other: Low nicotine content vape with tobacco e-liquids — Participants are randomly assigned to the order of each marketplace Group
  Arms: Low nicotine content vape with tobacco e-liquids

SUMMARY:
This study is proposing a four condition Electronic Tobacco Marketplace (ETM) study to determine if banning normal nicotine content (NNC) is sufficient for encouraging smokers to switch to potentially less harmful products or if the availability of higher nicotine and/or flavored alternative products (specifically e-cigarettes) are needed to achieve maximal reductions in smoking.

DETAILED DESCRIPTION:
The Family Smoking Prevention and Tobacco Control Act (FSPTCA) passed in 2009 provides the FDA with the authority to regulate tobacco products. One provision in this legislative act empowers the FDA to set limits on constituents in tobacco products, including nicotine. Such a measure has the potential to reduce the chance of individuals experimenting with smoking from becoming dependent and enable current smokers to quit when they are motivated to do so. Although the proposal to reduce nicotine in cigarettes has been met with skepticism by some because of concerns over compensatory smoking behavior and the potential emergence of a black market, this policy measure was considered to be technically feasible by the American Medical Association and the British Medical, by tobacco control researchers, policymakers and governmental officials who were convened in a meeting on nicotine regulation8, and by the World Health Organization Study Group on Tobacco Product Regulation. Most importantly, in July 2017, FDA Commissioner Gottlieb announced he was "directing our Center for Tobacco Products to develop a comprehensive nicotine regulatory plan premised on the need to confront and alter cigarette addiction." This announcement was followed on March 16, 2018 by the release of the Advance Notice of Proposed Rulemaking entitled "Tobacco Product Standard for Nicotine Level of Combusted Cigarettes" (ID: FDA-2017-N-6189-0001) "to obtain information for consideration in developing a tobacco product standard to set the maximum nicotine level for cigarettes."

This study proposes to conduct a within-subjects, multi-session virtual lab study and validation field assessment to determine how the availability of flavored e-liquids affects product purchasing among cigarette smokers. Adult daily cigarette smokers (N=64) will be recruited for this study. After initial eligibility is assessed, participants will complete six virtual sessions (1 baseline, 4 experimental, and 1 follow-up) and one field assessment to evaluate their tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years of age
* Self-report smoking at least 5 cigarettes per day for the past year
* Breathe carbon monoxide (CO) level > 8 ppm or positive urine NicCheck
* Willingness to use other tobacco products during the study
* Speak, comprehend, and read English sufficiently to complete study procedures
* Have home access to a computer, smart phone, or tablet with a web camera and internet access
* Tried a vaping device at least once in their lifetime

Exclusion Criteria:

* Currently seeking treatment to quit smoking
* Self-reported serious medical or psychiatric condition(s) including cardiovascular and chronic respiratory diseases
* Body temperature > 100.4 F
* Cold, flu or COVID-19 symptoms including fever, cough, and runny nose in the past 30 days
* Currently pregnant, breastfeeding or intending to become pregnant for the duration of the study or unwilling to agree to use adequate protection to avoid pregnancy
* CO reading > 80 ppm

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Donny, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarvis MJ, Bates C. Eliminating nicotine in cigarettes. Tob Control. 1999 Spring;8(1):106-7; author reply 107-9. No abstract available. PMID 10465828
- [Background] Kozlowski LT. Prospects for a nicotine-reduction strategy in the cigarette endgame: Alternative tobacco harm reduction scenarios. Int J Drug Policy. 2015 Jun;26(6):543-7. doi: 10.1016/j.drugpo.2015.02.001. Epub 2015 Feb 23. PMID 25795345
- [Background] Kozlowski LT. Cigarette prohibition and the need for more prior testing of the WHO TobReg's global nicotine-reduction strategy. Tob Control. 2017 Mar;26(e1):e31-e34. doi: 10.1136/tobaccocontrol-2016-052995. Epub 2016 Jun 29. No abstract available. PMID 27357937
- [Background] Kozlowski LT. Let actual markets help assess the worth of optional very-low-nicotine cigarettes before deciding on mandatory regulations. Addiction. 2017 Jan;112(1):3-5. doi: 10.1111/add.13515. Epub 2016 Aug 23. No abstract available. PMID 27554993
- [Background] Shatenstein S. Eliminating nicotine in cigarettes. Tob Control. 1999 Spring;8(1):106; author reply 107-9. No abstract available. PMID 10465827
- [Background] Henningfield JE, Benowitz NL, Slade J, Houston TP, Davis RM, Deitchman SD. Reducing the addictiveness of cigarettes. Council on Scientific Affairs, American Medical Association. Tob Control. 1998 Autumn;7(3):281-93. doi: 10.1136/tc.7.3.281. PMID 9825424
- [Background] Hatsukami DK, Perkins KA, Lesage MG, Ashley DL, Henningfield JE, Benowitz NL, Backinger CL, Zeller M. Nicotine reduction revisited: science and future directions. Tob Control. 2010 Oct;19(5):e1-10. doi: 10.1136/tc.2009.035584. PMID 20876072
- [Background] World Health Organization. WHO STUDY GROUP ON TOBACCO PRODUCT REGULATION. Report on the Scientific Basis of Tobacco Product Regulations: Fifth Report of a WHO Study Group. World Health Organ Tech Rep Ser. 2015;(989):1-234, back cover. PMID 26353746

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the initial 69 participants enrolled, 5 people were lost to follow up or withdrew between screening eligible and getting randomized to a group leaving 64 participants randomized. Staff instructed participants that one iteration of the task would be randomly selected and would determine which products (flavor e-liquids or tobacco e-liquids) they would use during the assessment. In reality, participants were only randomly assigned to tobacco e-liquid and never assigned to flavor e-liquid.
Period: Overall Study
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Started | 0 | 32 | 0 | 32
Completed | 0 | 29 | 0 | 32
Not Completed | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants that completed all virtual shopping trips before randomization of take-home products. Participants were told they may have a chance of taking home "all flavor e-liquids" to prevent purchasing bias, but they were only able to take home tobacco e-liquids.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids | Total
Number analyzed (Participants) | 0 | 32 | 0 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 |  | 0 | 0
  Between 18 and 65 years |  | 32 |  | 29 | 61
  >=65 years |  | 0 |  | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 49.2 (9.9) |  | 50.3 (12.6) | 50.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 18 |  | 18 | 36
  Male |  | 14 |  | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 4 | 4
  Not Hispanic or Latino |  | 32 |  | 28 | 60
  Unknown or Not Reported |  | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 1 |  | 1 | 2
  Asian |  | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0 | 0
  Black or African American |  | 16 |  | 15 | 31
  White |  | 15 |  | 16 | 31
  More than one race |  | 0 |  | 0 | 0
  Unknown or Not Reported |  | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 32 |  | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Purchased
Description: Average number of cigarettes purchased (analyzed as raw data and using derived behavioral economic measures)
Time Frame: Visit 6 approximately 4 weeks after baseline
Population: Among those participants who purchased cigarettes in Shopping Trip 7 at Virtual Visit 6, the average number of cigarettes purchased (in an experimental tobacco marketplace where packs of very low nicotine content (VLNC) cigarettes, bottles of e-liquid matched to their randomization condition, boxes of nicotine gum were available).
Measure: Mean (Standard Deviation); unit: average number of cigarettes
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
average number of cigarettes |  | 154.7 (131.7) |  | 119.2 (55.5)

2. Secondary Outcome: Number of E-liquid Milliliters Purchased
Description: Average number of e-liquid milliliters purchased (analyzed as raw data and using derived behavioral economic measures)
Time Frame: Visit 6 approximately 4 weeks after baseline
Population: Among those participants who purchased e-liquid in Shopping Trip 7 at Virtual Visit 6, the average number of mls purchased (in an experimental tobacco marketplace where packs of VLNC cigarettes, bottles of e-liquid matched to their randomization condition, boxes of nicotine gum were available).
Measure: Mean (Standard Deviation); unit: average number of milliliters
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
average number of milliliters |  | 36.7 (24.1) |  | 35.0 (29.6)

3. Secondary Outcome: Proportion of Participants Completing Flavor and Nicotine Content Discrete Choice Projections
Description: The proportion of participants projected to choose a cigarette over an e-cigarette under different potential regulatory scenarios, as determined by regression analysis.
Time Frame: Month 1 after baseline
Population: Scores reveal how important each product characteristic is to a participant when indicating their preference for one product over another (0 to 100, summing to 100). In our study, product type (2 levels: cigarette or e-cigarette), cigarette nicotine content (2 levels: normal or very low), e-liquid nicotine content (2 levels: 25mg/ml or 50mg/g) and available e-liquid flavor (2 levels: mint, fruit, sweet, tobacco or only tobacco) were manipulated in the discrete choice experiment.
Measure: Number; unit: Proportion of participants
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
Proportion of participants |  | 41.8 |  | 61.9

4. Secondary Outcome: Lung Cancer Perceived Risk Scores for VLNC Cigarettes
Description: The response options rely on a 10-point Likert-like scale: 1 = very low risk of disease; 2, 3, 4, 5, 6, 7, 8, 9, 10 = very high risk of disease. Minimum possible response 1. Maximum possible response 10. The higher the score, the greater perceived risk of VLNC cigarettes for lung cancer.
Time Frame: Baseline
Population: Group average for responses using a 10-point Likert-like scale: 1 = very low risk of disease; 2, 3, 4, 5, 6, 7, 8, 9, 10 = very high risk of disease. Minimum possible response 1. Maximum possible response 10. The higher the score, the greater perceived risk of VLNC cigarettes for lung cancer.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
score on a scale |  | 5.4 (2.9) |  | 4.2 (2.9)

5. Secondary Outcome: Product Evaluation Scale Scores
Description: Product evaluation scale scores for VLNC cigarettes among participants who received VLNC cigarettes will be determined by a product evaluation questionnaire. The questionnaire measures the strength of self-reported positive subjective effects (e.g., reward, satisfaction) following product use. The response options rely on a 7-point Likert-like scale: 1=not at all; 2= very little; 3= a little; 4= moderately; 5= a lot; 6= quite a lot; 7= extremely. The summed score adds responses to 13 separate items. Minimum possible response: 13. Maximum possible response: 91. Higher scores denote more favorable product effects. Note: This was only administered (at Virtual Visit 6) to participants who received each product type in the field (dependent on their baseline ETM shopping trip purchases).
Time Frame: Visit 6 approximately 4 weeks after baseline
Population: Group Averages, summed score of 13 items The product evaluation questionnaire measures the strength of self-reported positive effects (e.g., reward, satisfaction) following product use. The response options rely on a 7-point Likert-like scale: 1=not at all; 2= very little; 3= a little; 4= moderately; 5= a lot; 6= quite a lot; 7= extremely. Only administered to participants who received each product type in the field.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 19 | 0 | 30
score on a scale |  | 29.1 (15.3) |  | 29.1 (17.0)

6. Secondary Outcome: Minnesota Nicotine Withdrawal Scale Scores
Description: Minnesota Nicotine Withdrawal Scale measures the severity of nicotine withdrawal symptoms. The response options rely on a 5-point Likert-like scale; 0=None; 1= Slight; 2=Mild; 3=Moderate; 4=Severe. There are 7 items total, that are summed. Minimum possible response: 0. Maximum possible response: 28. Higher scores denote greater severity of withdrawal symptoms.
Time Frame: Visit 6 approximately 4 weeks after baseline
Population: Group averages, summed score of 7 items Minnesota Nicotine Withdrawal Scale measures the severity of nicotine withdrawal symptoms. The response options rely on a 5-point Likert-like scale; 0=None; 1= Slight; 2=Mild; 3=Moderate; 4=Severe. Minimum possible response: 0. Maximum possible response: 28. Higher scores denote greater severity of withdrawal symptoms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
score on a scale |  | 5.3 (5.9) |  | 4.9 (7.0)

7. Secondary Outcome: Questionnaire on Smoking Urges Score
Description: Questionnaire on Smoking Urges measures the strength of urges to smoke. The response options rely on a 7-point Likert-like scale: 1=Strongly Disagree; 2; 3; 4; 5; 6; 7= Strongly Agree. The questionnaire has 10 total items; scores sum responses to each item. Minimum possible response: 10. Maximum possible response: 70. Higher scores denote greater urges to smoke.
Time Frame: Visit 6 approximately 4 weeks after baseline
Population: Group averages, summed score of 10 items Questionnaire on Smoking Urges measures the strength of urges to smoke. The response options rely on a 7-point Likert-like scale: 1=Strongly Disagree; 2; 3; 4; 5; 6; 7= Strongly Agree. The questionnaire has 10 total items; scores sum responses to each item. Minimum possible response: 10. Maximum possible response: 70. Higher scores denote greater urges to smoke.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
score on a scale |  | 36.1 (18.7) |  | 32.4 (19.2)

8. Secondary Outcome: Tobacco Product Interest Scores
Description: Tobacco Product Interest of different products; Slider scale ranging from 0=No Interest to 100=Very Interested
Time Frame: 1 month after baseline
Population: Product interest toward different cigarettes and e-cigarettes; Slider scale ranging from 0 = No Interest to 100 = Very Interested
  Ppts were not actually randomized to "all flavor e-liquids"
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
score on a scale
  UB Cigs |  | 87.2 [0 to 100] |  | 88.4 [0 to 100]
  VLNC |  | 27.1 [0 to 100] |  | 32.2 [0 to 100]
  Pod E-Cig |  | 38.3 [0 to 100] |  | 33.2 [0 to 100]
  Mod E-Cig |  | 15.4 [0 to 100] |  | 35.6 [0 to 100]
  Pen E-Cig |  | 31.0 [0 to 100] |  | 40.3 [0 to 100]

9. Secondary Outcome: Tobacco Policy Questionnaire Scores
Description: Tobacco Policy Questionnaire scored from Support, Oppose, and Don't know for personal opinions on Making Cigarettes Less Addictive
Time Frame: 1 month after baseline
Population: Ppts were not actually randomized to "all flavor" e-liquid groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
Number analyzed (Participants) | 0 | 29 | 0 | 32
Participants
  Support |  | 15 |  | 11
  Oppose |  | 7 |  | 11
  Don't Know |  | 7 |  | 10

10. Other Pre Specified Outcome: Product Use Themes Emerging From the Qualitative Interviews
Description: Participants are asked about their opinions and experiences using tobacco products other than their usual brand during the field assessment.
Time Frame: Screening visit through end of study (up to week eight)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Tobacco Product Use During Field Assessment
Description: Participants are asked what products they had used and quantity every day during the field assessment.
Time Frame: Screening visit through end of study (up to week eight)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Biomarkers of Exposure During Field Assessment - Carbon Monoxide
Description: Product use and biomarkers of exposure during the field assessment will be analyzed using linear regression or other appropriate regression models. The model for primary analysis of these data will include main effects for each of the two factors (for the ETM condition carried into the field assessment), and the corresponding baseline measure to improve precision. Carbon Monoxide (CO) is collected in ppm.
Time Frame: Screening visit through end of study (up to week eight)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Biomarkers of Exposure During Field Assessment - Cotinine
Description: Product use and biomarkers of exposure during the field assessment will be analyzed using linear regression or other appropriate regression models. The model for primary analysis of these data will include main effects for each of the two factors (for the ETM condition carried into the field assessment), and the corresponding baseline measure to improve precision. Cotinine is collected in ng/ml.
Time Frame: Screening visit through end of study (up to week eight)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Screening visit through end of study (up to week eight)
Description: Number of participants at risk is zero for two of the groups because no participants were assigned to those groups.
Arm/Group | Normal Nicotine Content Vape With All Flavor E-liquids | Normal Nicotine Content Vape With Tobacco E-liquids | Low Nicotine Content Vape With All Flavor E-liquids | Low Nicotine Content Vape With Tobacco E-liquids
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/29 | 0/0 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/29 | 0/0 | 0/32
Other Adverse Events (participants affected / at risk) | 0/0 | 1/29 | 0/0 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Nicotine Content Vape With All Flavor E-liquids (N=0) | Normal Nicotine Content Vape With Tobacco E-liquids (N=29) | Low Nicotine Content Vape With All Flavor E-liquids (N=0) | Low Nicotine Content Vape With Tobacco E-liquids (N=32)
Stress/Irritability (Psychiatric disorders) | 0 | 1 (1) | 0 | 1 (1) — Two Participants experienced an increase in stress; due to the lower nicotine amount in cigs they reported.
COVID (Infections and infestations) | 0 | 0 (0) | 0 | 1 (1) — Tested positive for COVID during trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT05320887/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05320887/ICF_000.pdf